CLINICAL TRIAL: NCT03621839
Title: New Diagnosis or Prognosis Biomarkers for Alzheimer's Disease: Biobank of CSF Collected as Part of Differential Diagnosis of Dementia
Brief Title: New CSF Biomarkers for Alzheimer's Disease
Acronym: BioAD
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Catherine MALAPLATE, MCU-PH, Central Hospital, Nancy, France
Other Study IDs: 2012-PSS/COLL- LCR/ARMAND/MS
Record Dates: First submitted 2018-07-25; First posted 2018-08-09 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Dementia; Neurodegenerative Diseases
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Today, the Alzheimer's disease (AD) diagnosis is founded not only on clinical criteria but also on complementary examinations to confirm a physiopathological process of AD. In complex cases, lumbar punction could be necessary in order to measure Aβ peptides and Total and phosphorylated Tau but new biomarkers could be useful. The main objective of this project is to conserve these cerebrospinal fluids, collected in usual practice in order to validate new biomarkers for diagnosis, prognosis or therapeutic following of Alzheimer's disease and other dementia.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar punction collected in usual practice in the context of dementia diagnosis

Exclusion Criteria:

* Absence of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consenting patients submitted to a lumbar punction in the context of dementia diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2013-07-12 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
CSF collection constitution to have samples available for assessing new Alzheimer's biomarker | 50 years
  Each CSF collected in the context of dementia diagnosis were conserved to be used in other studies on Alzheimer's or dementia biomarkers. Futre studies that will use collected CSF to assess new biomarkers will be conduced under a new protocol describing scientific contexte, specific aims and time frame necessary to achieve them.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU De Nancy, Nancy, Grand Est, France